CLINICAL TRIAL: NCT04113798
Title: Exercise and Therapeutic Learning Among Women With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0845; A538900 (Other: UW Madison); SMPH/PSYCHIATRY/PSYCHIATRY (Other: UW Madison); Protocol Version 11/4/2019 (Other: UW Madison)
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: PTSD
Keywords: women; exercise; mental health
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Intensity Exercise (Experimental): Day 1 Assessment, Day 2 Fear Learning, Day 3 Fear Extinction (followed by moderate intensity exercise), Day 4 Recall of Fear Extinction
  Interventions: Other: Day 1 Assessments; Other: Day 2 Fear Learning; Other: Day 3 Fear Extinction; Behavioral: Moderate Intensity Exercise; Other: Day 4 Recall of Fear Extinction
- Control (Active Comparator): Day 1 Assessment, Day 2 Fear Learning, Day 3 Fear Extinction (followed by low intensity exercise), Day 4 Recall of Fear Extinction
  Interventions: Other: Day 1 Assessments; Other: Day 2 Fear Learning; Other: Day 3 Fear Extinction; Behavioral: Low Intensity Exercise; Other: Day 4 Recall of Fear Extinction

INTERVENTIONS:
Other: Day 1 Assessments — Structured clinical interview to assess trauma history and mental health diagnoses, as well as a screening EKG to assess safety to engage in exercise testing (lasts 3-4 hours)
Other: Day 2 Fear Learning — Participants undergo a standard fear conditioning procedure, in which they learn that one of two geometric shapes (circles or triangles) predict the occurrence of a noxious stimulus (mild electrotactile stimulation). Day 2 lasts about 1 hour.
Other: Day 3 Fear Extinction — Participants undergo a fear extinction procedure, in which participants learn that the geometric shapes no longer predict a noxious stimulus (i.e., safety learning). Blood samples will be drawn immediately before exercise, and immediately following.
Behavioral: Moderate Intensity Exercise — The moderate-intensity aerobic exercise session will consist of a 5 minute warm-up of light intensity activity (40-60% maximum heart rate; MHR) on a treadmill followed by walking or running at a moderate intensity (i.e., between 70-75% MHR) for 30 minutes on Day 3
  Arms: Moderate Intensity Exercise
Behavioral: Low Intensity Exercise — Control participants will maintain light-intensity activity (i.e., walking at ~50% of MHR) for the full duration of 30 minutes.
  Arms: Control
Other: Day 4 Recall of Fear Extinction — During Day 4, recall of the fear extinction memory is tested. Visits on Day 4 occur ~24 hours following Day 3, and lasts about 30 minutes.

SUMMARY:
This study aims to test whether aerobic exercise performed after fear extinction learning improves the consolidation and subsequent recall of the learned safety memories (i.e., fear extinction memories) among adult women with PTSD related to interpersonal violence exposure, and whether this effect is mediated by the ability of exercise to increase acute levels of Brain-Derived Neurotrophic Factor (BDNF) and endocannabinoids (eCB). Participants can expect to be on study for up to 90 days, participating in 4 study stages: Day 1 of Assessments, Day 2 of Fear Learning, Day 3 of Fear Extinction (and activity), and Day 4 of Recall of Fear Extinction.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of PTSD where the index traumatic event includes physical or sexual assault
* English speaking
* Medically healthy

Exclusion Criteria:

* Any endorsed medical concerns related to physical activity (as probed in the phone screening questions regarding cardiovascular, pulmonary, or metabolic disease and as assessed via the Physical Activity Readiness Questionnaire (PAR-Q), which probes into participants' history of heart conditions, chest pain, dizziness, loss of consciousness, bone/joint problems, and medication history). Participants would not be excluded if they report this condition being "controlled" or "addressed" through medication or lifestyle change, such as regular exercise.
* Major medical disorders (such as cancer, AIDS)
* Physical discomfort or difficulty with blood draws
* Psychotic disorders
* Intellectual disabilities
* Developmental disorders
* Active substance use disorders
* Pregnancy
* Due to safety concerns, participants with these conditions will be ineligible to participate:

  * Major medical disorders (e.g., HIV, cancer)
  * Daily cannabis use
  * History of light headedness or fainting during blood draws or physical activity
  * History of chest pain during physical activity
  * Abnormal EKG finding at intake visit screening, without follow-up clearance from their physician
  * Bone, joint, cardiac, pulmonary, metabolic, or other medical conditions that may be worsened by physical activity (e.g., Chronic Obstructive Pulmonary Disease (COPD), diabetes, hypertension) that is not currently addressed via medication or lifestyle change.
  * A positive pregnancy test
  * A self-reported history of loss of consciousness (greater than 30 minutes)
  * Physical disabilities that prohibit task performance (such as blindness or deafness)
  * Psychotic disorders (e.g., schizophrenia)
  * Any other condition that the investigator believes might put the participant at risk

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 35 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Participant Skin Conductance Responding (SCR) | up to Day 4
  Aim 1 fear extinction analyses consists of a 2 (group: low-intensity exercise vs moderate-intensity exercise) x 2 (cue: conditioned fear and safety) x 2 (task phase context: learning context vs extinction context) mixed design focused on Day 4 fear responding (skin conductance responses). SCR data will be acquired on a BIOPAC MP150 Data Acquisition System (BIOPAC Systems, Inc.) with electrodes placed on participant's left hand. Participants will be instructed to select an intensity of a 7/10 on the subjective pain scale, which should be "uncomfortable, but not painful." Average intensity of participant skin conductance will be reported.
Group Differences in Serum Brain-Derived Neurotrophic Factor (BDNF) | before and after 30 min exercise on Day 3
  Aim 2 group differences in BDNF consists of a 2 (group: moderate-intensity vs low-intensity) x 2 (cue: conditioned fear and safety) x 2 (task phase context: learning context vs extinction context) x 2 (timepoint: pre condition vs post condition,) mixed design. The hypothesis is BDNF increases following exercise will separately mediate the relationship between aerobic exercise and enhanced fear extinction recall.
Group Differences in Serum Endocannabinoid (eCB) Content | before and after 30 min exercise on Day 3
  Aim 2 group differences in eCB consists of a 2 (group: moderate-intensity vs low-intensity) x 2 (cue: conditioned fear and safety) x 2 (task phase context: learning context vs extinction context) x 2 (timepoint: pre condition vs post condition,) mixed design. The hypothesis is eCBs increases following exercise will separately mediate the relationship between aerobic exercise and enhanced fear extinction recall.

SECONDARY OUTCOMES:
Change in Profile of Mood States (POMS) Questionnaire | at each visit, up to Day 4
  The POMS survey is a 65-item survey scored on a 5 point Likert Scale (0-4) where 0 s 'not at all' and 4 is 'extremely' for the tension, depression, fatigue, confusion, and anger subscales, and reversed for the vigor and esteem-related affect subscales. The range of total possible scores is XX-XX with higher numbers indicating more extreme or negative moods.
Change in State-Trait Anxiety Inventory (STAI) | at each visit, up to Day 4
  STAI is a 20-item assessment rated on a 4-point scale from 'almost never' to 'almost always' with the total scores ranging from 20-80. Higher scores indicate greater anxiety.
Change in Positive and Negative Affect Scale (PANAS) | at each visit, up to Day 4
  PANAS is comprised of two 10-item scales for both positive and negative affect. Total combine scoring is from 20-100 where the higher the score the more negative the affect.

CONTACTS AND LOCATIONS:
Overall Officials: Josh Cisler, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crombie KM, Sartin-Tarm A, Sellnow K, Ahrenholtz R, Lee S, Matalamaki M, Adams TG, Cisler JM. Aerobic exercise and consolidation of fear extinction learning among women with posttraumatic stress disorder. Behav Res Ther. 2021 Jul;142:103867. doi: 10.1016/j.brat.2021.103867. Epub 2021 Apr 27. PMID 34020153